CLINICAL TRIAL: NCT01501500
Title: Therapeutic Effect of Botulinum Toxin Type A in Addition to Total Contact Insole in Treating Painful Hallux valgus-a Pilot Study
Brief Title: Effect of Botulinum Toxin to Hallux Valgus in Addition to Total Contact Insole
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSC 99-2314-B-182A-020
Record Dates: First submitted 2011-12-21; First posted 2011-12-29 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2010-03

CONDITIONS: Hallux Valgus
Keywords: botulinum toxin type A; hallux valgus angle; foot function index; VAS pain scale
MeSH Terms: conditions — Hallux Valgus | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- botulinum toxin type A. HV angle (Active Comparator): intramuscular injection of BTA into target muscle
  Interventions: Drug: BOTOX
- Normal saline, HV angle (Placebo Comparator): intramuscular injection of normal saline into target muscle
  Interventions: Drug: Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: BOTOX — once injection of BTA 3oU into hallux oblique and transverse heads each
  Other Names: BOTOX (Allergan, Irvine, CA)
  Arms: botulinum toxin type A. HV angle
Drug: Normal Saline (0.9% NaCl) — Normal saline 0.3ml to oblique and transverse heads each
  Arms: Normal saline, HV angle

SUMMARY:
The investigators propose a new therapeutic approach by injecting Botulinum Toxin Type A (BTA) to the oblique and transverse heads of adductor muscle of the great toe. BTA works by binding presynaptically to high-affinity recognition sites on the cholinergic nerve terminals and decrease the release of acetylcholine, causing a neuromuscular blocking effect. The investigators hypothesize that BTA injection may help to decrease the hallux valgus angle by decrease adductor hallucis muscle activation. Thereby enhance the therapeutic result of hallux valgus treated with total contact insole. The outcome measurement may shed light in treating patient with painful hallux valgus and document evidence for plantar pressure changes in acute, sub-acute and chronic stage.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled prospective study to assess the influence and efficacy of intramuscular (IM) Botulinum Toxin Type A (BTA) injection in patients with painful hallux valgus with the use of total contact insole.

Fifty feet with painful hallux valgus will be collected. Informed consent is obtained according to the hospital's medical ethics and the human clinical trial committee. The feet will be randomized into 2 groups: Group A (n=25, treatment group) and Group B (n=25, control group). Clinical diagnosis of hallux valgus is made based on observation of great toe lateral deviation. Inclusion criteria were hallux valgus with angle of at least 20°, single or bilateral hallux valgus. To obtain the hallux valgus angle, foot roentgenography in AP and sesamoid views under the weight bearing condition will be obtained. The angle formed by lines drawn to bisect the first metatarsal bone and the proximal phalanx of the great toe will be measured. The exclusion criteria include history of foot operations, rheumatoid and gouty arthritis, and any contraindication to BTA administration. Subjective data such as the Foot Function Index will be collected.

ELIGIBILITY:
Inclusion Criteria:

* hallux valgus with angle of at least 20°,
* single or bilateral hallux valgus.

Exclusion Criteria:

* history of foot operations,
* rheumatoid arthritis and gouty arthritis.
* Any contraindication on BTA administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
hallux valgus angle | up to 18 months
  radiological assessment before and after the intervention

SECONDARY OUTCOMES:
foot function index for quality of life | up to 18 months
  Foot Function Index before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Katie P Wu, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung MH, Guishan, Taoyuan, Taiwan

REFERENCES:
- [Derived] Wu KP, Chen CK, Lin SC, Pei YC, Lin RH, Tsai WC, Fuk-Tan Tang S. Botulinum Toxin type A injections for patients with painful hallux valgus: a double-blind, randomized controlled study. Clin Neurol Neurosurg. 2015 Feb;129 Suppl 1:S58-62. doi: 10.1016/S0303-8467(15)30014-7. PMID 25683315